CLINICAL TRIAL: NCT02402985
Title: Comparison of a High-protein, Carbohydrate-restricted Diet With a High Proportion of Leguminous Protein Compared to Animal Protein on Metabolic Control in Patients With Type 2 Diabetes, "LeguAN Study"
Brief Title: Comparison of a Plant Protein Diet to a Animal Protein Diet Emphasized in Type 2 Diabetics
Acronym: LeguAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: Ministry of Food and Agriculture, Germany (Unknown); Ernst von Bergmann Hospital (Other); University Hospital Tuebingen (Other); Institute of Gain Processing IGV GmbH, Potsdam (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Director/Dep. Clinical Nutrition, German Institute of Human Nutrition
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BMLEV-Project
Record Dates: First submitted 2015-02-04; First posted 2015-03-31 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus, Type 2; Nutrition Disorders; Obesity; Body Weight; Metabolic Syndrome x; Metabolic Diseases
Keywords: nutritional support; diet therapy; protein diet; isocaloric diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Nutrition Disorders; Obesity; Body Weight; Metabolic Syndrome; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High animal protein diet group AP (Other): 6-weeks diet intervention with high animal protein
  Interventions: Other: High animal protein diet group
- High plant protein diet group PP (Other): 6-weeks diet intervention with high plant protein
  Interventions: Other: High plant protein diet group

INTERVENTIONS:
Other: High animal protein diet group — 25-30% protein, 40 % carbohydrates, 30-35 % fat over 6 weeks
  Arms: High animal protein diet group AP
Other: High plant protein diet group — 25-30% protein, 40 % carbohydrates, 30-35 % fat over 6 weeks
  Arms: High plant protein diet group PP

SUMMARY:
This 6-week parallel randomised prospective dietary intervention study with type 2 Diabetes investigates the nutrition influence of animal protein in comparison to plant protein on the glucose metabolism.

DETAILED DESCRIPTION:
2x20 patients with Diabetes mellitus type 2 are randomise by a blind computer assist for an equal allocation in both groups (animal protein vs. plant protein). The food components for both groups are 40% carbohydrates, 30% fat and 30% protein. The carbohydrates are correspond with a high fiber content and a low blood sugar effectiveness of carbohydrates (glycemic index).

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus, type 2
* HbA1c between 6-11%

Exclusion Criteria:

* Consumptive or high grade diseases
* Intake of metabolic influence a/o anticoagulent drugs (e.g. cortisone, ASS, antibiotics)
* Diabetes type 1
* Pregnancy
* Chronic disease of heart, kidney, liver
* High grade anaemia
* High grade infection disease
* Relevant change of body weight (+/- 5 kg) since 8 weeks before begin of study Intervention
* Missing data about primary outcome measures (hyperinsulinaemic euglycaemic clamp, mealtime test, data about dietary intake from food diaries or food protocols)
* Significant deviation from dietary targets during the monitored 6 weeks isoenergetic period
* Allergies including food allergies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Variance of glucose metabolism after different diet intervention | week 0 and 6
  Change of insulin sensitivity measured by hyperinsulinaemic euglycaemic clamp and meal time test (MTT)

SECONDARY OUTCOMES:
Development of indices for the prediction of liver fat mass | week 0 and 6
  Change of fat fraction in liver, abdominal and in the total body fat measuring by MRI/H1-spectroscopy
Development of indices for the prediction of body fat mass | week 0, 2, 4 and 6
  Change of body fat measuring by body composition assessment (BODPOD) and bioelectrical impedance analysis (BIA)
Expression Change of inflammatory markers in blood and fat tissue | week 0 and 6
  Measurement of gene expression of inflammation cytokines
Modification of epigenetic DNA | week 0 and 6
Changes of gastrointestinal microbiota | week 0 and 6
  Molecular mechanisms between nutrition, intestinal bacteria and host
Variance of composite biometric data | week 0, 2, 4 and 6
  Change of blood pressure, weight, body mass index, waist-hip ratio
Variance of blood data | week 0, 2, 4 and 6
  Changes in the levels of composite circulating inflammatory and metabolic syndrome biomarkers
Variance of intestinal hormones | week o and 6
  Change of intestinal hormones measured with a meal time test (MTT)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas FH Pfeiffer, Prof, Principal Investigator — German Institute of Human Nutrition, Potsdam-Rehbrücke, Nuthetal, Germany
Locations (1):
- German Institute of Human Nutrition, Potsdam-Rehbruecke, Nuthetal, Germany

REFERENCES:
- [Derived] Kabisch S, Markova M, Hornemann S, Sucher S, Pivovarova-Ramich O, Machann J, Hierholzer J, Rohn S, Pfeiffer AFH. Liver fat scores do not reflect interventional changes in liver fat content induced by high-protein diets. Sci Rep. 2021 Apr 23;11(1):8843. doi: 10.1038/s41598-021-87360-2. PMID 33893355
- [Derived] Markova M, Koelman L, Hornemann S, Pivovarova O, Sucher S, Machann J, Rudovich N, Thomann R, Schneeweiss R, Rohn S, Pfeiffer AFH, Aleksandrova K. Effects of plant and animal high protein diets on immune-inflammatory biomarkers: A 6-week intervention trial. Clin Nutr. 2020 Mar;39(3):862-869. doi: 10.1016/j.clnu.2019.03.019. Epub 2019 Mar 27. PMID 30967307
- [Derived] Markova M, Hornemann S, Sucher S, Wegner K, Pivovarova O, Rudovich N, Thomann R, Schneeweiss R, Rohn S, Pfeiffer AFH. Rate of appearance of amino acids after a meal regulates insulin and glucagon secretion in patients with type 2 diabetes: a randomized clinical trial. Am J Clin Nutr. 2018 Aug 1;108(2):279-291. doi: 10.1093/ajcn/nqy100. PMID 29982277
- [Derived] Markova M, Pivovarova O, Hornemann S, Sucher S, Frahnow T, Wegner K, Machann J, Petzke KJ, Hierholzer J, Lichtinghagen R, Herder C, Carstensen-Kirberg M, Roden M, Rudovich N, Klaus S, Thomann R, Schneeweiss R, Rohn S, Pfeiffer AF. Isocaloric Diets High in Animal or Plant Protein Reduce Liver Fat and Inflammation in Individuals With Type 2 Diabetes. Gastroenterology. 2017 Feb;152(3):571-585.e8. doi: 10.1053/j.gastro.2016.10.007. Epub 2016 Oct 17. PMID 27765690